CLINICAL TRIAL: NCT06437444
Title: Asthma Crisis in Paediatrics: Impact of a Care Pathway in Primary and Hospital Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Basque Health Service (Other Government)
Collaborators: Health Department of the Basque Government (Unknown)
Responsible Party: Principal Investigator, Marta Montejo Fernandez, Principal Investigator, Basque Health Service
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021111010
Record Dates: First submitted 2024-05-26; First posted 2024-05-31 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Asthma in Children; Implementation Science

STUDY DESIGN:
Intervention Model Description: Quasi-experimental pre-post cluster trial with control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Asthma Care Pathway group (Experimental): All the primary care and hospital pediatricians of the two Integrated Hospital Organizations (IHO) (Barakaldo-Sestao and Ezkerraldea-Enkarterri-Cruces) where the care pathway will be implemented. 83 participants in total.
  Interventions: Behavioral: The implementation strategy to encourage the adoption of the Care Pathway
- Control (No Intervention): Primary care and hospital pediatricians of other IHOs where the care pathway is not implemented, but with similar characteristics to those in the experimental group, and with a proportion of 1:2. 166 participants in total.

INTERVENTIONS:
Behavioral: The implementation strategy to encourage the adoption of the Care Pathway — 1. Dissemination of the most novel aspects of the agreed Care Pathway via corporate mail.
  2. Integration of information and communication tools into electronic health records to facilitate the recording and the standardized implementation of recommended practice.
  3. Audit & Feedback (A&F) data reports, sent monthly, to each paediatrician on the rate of prescription of bronchodilators administered with a spacer chamber, together with the rates of the other indicators established in the pathway, in their health centre and in the rest of the centres in the participating health areas.
  4. Interactive training sessions, in which epidemiological data and data on the health, economic and social impact of asthma attacks were presented, together with data on other indicators associated with the care pathway, and key messages on current treatment recommendations based on the latest clinical practice.
  5. Distribution of reminder posters in paediatrics consultations, PEDs and health centers.
  Arms: Asthma Care Pathway group

SUMMARY:
This study aims to evaluate the effect of the implementation of the new Asthma Integrated Care Pathway in the Basque Healthcare Service for the improvement of care for children with asthma attacks and the reduction of variability between professionals and care settings in this care practice. Asthma is the most common chronic disease in children and has a major impact on people's quality of life. The Asthma Integrated Care Pathway is a structured multidisciplinary care plan that details the essential steps in the care of patients with mild-moderate asthma attacks and the coordinated practice of the agents involved as dictated by the evidence. This pathway will include quality indicators of compliance with diagnostic criteria, assessment of severity and prescription of drugs, as well as the experience of families and professionals, which have been collected in meetings designed for this purpose.

The study consists in a mixed methods implementation trial with two phases:

1. Phase I: a quantitative evaluation will be carried out to assess implementation outcomes at the professional level through a pretest-posttest quasi-experimental study with paired control group, with a ratio of 1:2. The primary outcome variable will be the overall percentage of bronchodilator treatment with a spacer chamber in children diagnosed with mild-moderate asthma attacks. We will also include as outcomes to be measured the registration rate of the Pulmonary Score, the recording rate of the assessment of persistent asthma symptoms, and the rate of initiation of background treatment in children with persistent asthma symptoms. These variables will be analysed using differences in pre- and post-intervention outcome measures between the intervention and control groups.
2. Phase II: a qualitative evaluation will be carried out through a structured process with discussion groups focused on the identification of the main barriers and facilitators for the provision of recommended clinical practice related to asthmatic crisis in mild-moderate cases established by the Asthma Integrated Care Pathway. A purposive sample of paediatricians stratified by level of care and service organisations will be recruited to ensure that all views are represented in the discussion groups. The structured script will be designed with questions to explore each of the domains of the Theoretical Domains Framework (TDF).

The study will be carried out mainly in two integrated healthcare organizations (IHO), which are made up of two primary care areas and the paediatric reference hospital emergency department of both areas, as well as the hospitalisation, intensive care and paediatric pneumology departments of said hospital, to extend in the future the Asthma Integrated Care Pathway to the rest of the Basque Health Service IHOs.

ELIGIBILITY:
Eligibility for professionals:

* Primary Care paediatricians and nurses
* Paediatricians and nurses in the Paediatric Emergency Department
* Paediatricians and nurses on the inpatient ward
* Paediatric Intensive Care paediatricians and nurses
* Paediatric Pneumology paediatricians and nurses

Eligibility for patients:

Patients between 2 and 14 years,that have being attended between the 7 May 2023 and the 7 May 2025, and with an acute episode of asthma, defined as:

* an episode of wheezing and a previous diagnosis of asthma or with a previous episode of wheezing
* a first episode in a child older than 2 years with a personal/family history of atopy and/or with an objective response to bronchodilators as assessed by the Pulmonary Score

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 249 (Estimated)
Dates: Start 2023-05-07 (Actual); Primary Completion 2026-05-07 (Estimated); Study Completion 2026-05-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of bronchodilator treatment | from baseline to 12 months, 24 months and 36 months
  The overall percentage of bronchodilator treatment with a spacer chamber in children diagnosed with mild-moderate asthma attacks.

SECONDARY OUTCOMES:
Pulmonary Score registration | from baseline to 12 months, 24 months and 36 months
  Rate of Pulmonary Score registration in children diagnosed with mild-moderate asthma attacks, at all levels of care.
Assessment and recording of persistent asthma symptoms. | from baseline to 12 months, 24 months and 36 months
  Rate of assessment and recording of persistent asthma symptoms in children diagnosed with mild-moderate asthma attacks by ussing the PACT form (Pediatric Asthma Control Tool).
Initiation of background treatment in children with persistent asthma symptoms | from baseline to 12 months, 24 months and 36 months
  Rate of initiation of background treatment in children who have been assessed and registered with persistent asthma symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Primary Care Research Unit of Bizkaia, Barakaldo, Bizkaia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared that underlie results reported in the publication, after deidentification.
Supporting Information: Study Protocol
Time Frame: Starting 6 months after the publication of results
Access Criteria: Since data supporting the present study will mostly concern routine data retrieved from the electronic health record of the Basque Health Service-Osakidetza, it will be only shared on justified request to the study guarantors (proposals should be directed to the Responsible Party). It will only be shared with researchers whose proposed use of the data has been approved by an independent review committee identified for this purpose.

REFERENCES:
- [Derived] Montejo M, Paniagua N, Sanchez A, Rueda-Etxebarria M, Pijoan JI, Saiz Hernando C, Martin V, Vazquez Ronco MA, Santiago Burruchaga M, Garcia Urabayen D, Perez Llarena G, Castelo S, Benito J. Improving the management of acute asthma in children through an integrated care pathway: an implementation study protocol. Front Pediatr. 2025 Aug 19;13:1646499. doi: 10.3389/fped.2025.1646499. eCollection 2025. PMID 40904739